CLINICAL TRIAL: NCT05250050
Title: Clinical Efficacy and Health Economic Evaluation of Susceptibility-Guided Therapy for Helicobacter Pylori Infection Treatment：Multicenter Randomized Controlled Study
Brief Title: Susceptibility-Guided Therapy for Helicobacter Pylori Infection Treatment
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B2021-831
Record Dates: First submitted 2022-02-11; First posted 2022-02-22 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Helicobacter Pylori Infection
MeSH Terms: interventions — Esomeprazole; Metronidazole; Clarithromycin; Levofloxacin; Amoxicillin; Tetracycline

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The technicians, who performed culture, antimicrobial susceptibility testing or urea breath test were blinded to treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Genotypic resistance guided therapy (Experimental): After Helicobacter pylori drug resistance mutation gene detection, according to genotypic antibiotic resistance pattern of each one, give esomeprazole 20mg bid and bismuth potassium citrate 0.6 g bid, combined two sensitive antibiotics of Amoxicillin, tetracycline,clarithromycin, metronidazole,and levofloxacin. All regimens will be given for 14 days.
  Interventions: Drug: Esomeprazole; Drug: Bismuth potassium citrate; Drug: Metronidazole; Drug: Clarithromycin; Drug: Levofloxacin; Drug: Amoxicillin; Drug: Tetracycline
- Phenotypic resistance guided therapy (Experimental): After antimicrobial susceptibility testing of Helicobacter pylori from biopsy samples, according to phenotypic antibiotic resistance pattern of each one, give esomeprazole 20mg bid and bismuth potassium citrate 0.6 g bid, combined two sensitive antibiotics of Amoxicillin, tetracycline,clarithromycin, metronidazole,and levofloxacin. All regimens will be given for 14 days.
  Interventions: Drug: Esomeprazole; Drug: Bismuth potassium citrate; Drug: Metronidazole; Drug: Clarithromycin; Drug: Levofloxacin; Drug: Amoxicillin; Drug: Tetracycline
- Empiric therapy (Active Comparator): Esomeprazole 20 mg bid, bismuth potassium citrate 0.6 g bid, metronidazole 0.4 g qid, and Amoxicillin 1.0 g bid (no penicillin allergy) OR tetracycline 0.5g qid (penicillin allergy) for 14 days
  Interventions: Drug: Esomeprazole; Drug: Bismuth potassium citrate; Drug: Metronidazole; Drug: Amoxicillin; Drug: Tetracycline

INTERVENTIONS:
Drug: Esomeprazole — 20mg bid
Drug: Bismuth potassium citrate — 0.6g bid
Drug: Metronidazole — 0.4g qid
Drug: Clarithromycin — 0.5g bid
  Arms: Genotypic resistance guided therapy; Phenotypic resistance guided therapy
Drug: Levofloxacin — 0.5g qd
  Arms: Genotypic resistance guided therapy; Phenotypic resistance guided therapy
Drug: Amoxicillin — 1g bid
Drug: Tetracycline — 0.5g qid

SUMMARY:
This multicenter randomized controlled clinical trial was conducted to compare the eradication efficacy and health economic benefits of individualized regimens based on HP drug resistance mutation gene detection (multiple PCR method), individualized regimens based on HP traditional drug sensitivity testing (E-test method) and empirical regimens in the Helicobacter pylori treatment.

DETAILED DESCRIPTION:
This multicenter randomized controlled clinical trial was conducted to compare the eradication efficacy and health economic benefits of individualized regimens based on HP drug resistance mutation gene detection (multiple PCR method), individualized regimens based on HP traditional drug sensitivity testing (E-test method) and empirical regimens in the treatment of Helicobacter pylori in patients with chronic gastritis. This study will compare the efficacy of individualized and empirical drug sensitivity regimens, and conduct cost-effectiveness analysis to provide pharmacoeconomic guidance for clinical decision-making. At the same time, it will provide reference for the reasonable pricing of H.pylori drug sensitivity test and considering the health benefits brought by its inclusion in medical insurance.

ELIGIBILITY:
Inclusion Criteria:

* Participate in the trial voluntarily, fully understand the trial, and sign the informed consent form (ICF).
* 18-75 years old on the day of signing the ICF.
* Helicobacter pylori infection confirmed by 13C-urea breath test or rapid urease test.

Exclusion Criteria:

* Patients with severe heart, lung, kidney, liver, blood, nerve, endocrine, and psychiatric diseases.
* Subjects or guardians refused to participate in the trial.
* Alcohol and/or drugs Abuse (addiction or dependence) or poor compliance with doctor's judgment.
* Have taken antibiotics, bismuth, proton pump inhibitors or Chinese traditional medicine 4 weeks before treatment.
* Pregnant or lactating women.
* Active peptic ulcer.
* allergic to drugs used in the trial.
* any other circumstances that are not suitable for recruitment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 388 (Estimated)
Dates: Start 2022-03-25 (Estimated); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Eradication rate of Helicobacter pylori | 6 weeks
  Eradication of Helicobacter pylori was defined as negative result of urea breath test (<4‰ cut-off value).

SECONDARY OUTCOMES:
Eradication rate of Helicobacter pylori resistant strains | 6 weeks
  Eradication of Helicobacter pylori was defined as negative result of urea breath test (<4‰ cut-off value). The antibiotic resistant strains were assessed using the E test method.
Eradication rate of Helicobacter pylori susceptible strains | 6 weeks
  Eradication of Helicobacter pylori was defined as negative result of urea breath test (<4‰ cut-off value). The antibiotic susceptible strains were assessed using the E test method.

OTHER OUTCOMES:
Adherence rate | 2 weeks during therapy
  The proportion of subjects with good adherence. Good adherence was defined as that subjects took more than 80% of the total medication.
Frequency of adverse events | 2 weeks during therapy
  Any possible adverse events during the 14-day treatment period were recorded.
Average cost of each group | 6 weeks
  Average medical cost related to therapy and followup in each group

CONTACTS AND LOCATIONS:
Overall Officials: Hong Gao, MD, Principal Investigator — Fudan University
Locations (3):
- China (3):
  - Renji Hospital, School of Medicine, Shanghai Jiaotong University, Shanghai, Shanghai Municipality
  - Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be available from the principal investigator Hong Gao at gao.hong@zs-hospital.sh.cn, beginning 6 months and ending 5 years after the trial results were published. The study protocol and statistical analysis plan are available online from https://clinicaltrials.gov/. All proposals requesting data access will need to specify how it is planned to use the data, and all proposals will need approval of all investigators before data release.
Supporting Information: Study Protocol
Time Frame: Beginning 6 months and ending 5 years after the trial results were published.
Access Criteria: All proposals requesting data access will need to specify how it is planned to use the data, and all proposals will need approval of all investigators before data release.
URL: http://clinicaltrials.gov/